CLINICAL TRIAL: NCT02510456
Title: Monitoring Neoadjuvant Chemotherapy Response In Breast Cancer Patients Using Diffuse Optical Spectroscopic Imaging (DOSI)
Brief Title: Monitoring Neoadjuvant Chemotherapy Response in Breast Cancer Patients Using Diffuse Optical Spectroscopic Imaging
Acronym: DOSI
Status: Completed | Type: Observational
Sponsor: Boston Medical Center (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: H-33188; RSG-14-015-01-CCE (Other Grant/Funding Number: American Cancer Society); DOSI (Other: Boston Medical Center)
Record Dates: First submitted 2015-03-09; First posted 2015-07-29 (Estimated); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer
Keywords: Diffuse Optical Spectroscopy Imaging (DOSI)
MeSH Terms: conditions — Breast Neoplasms | interventions — Cohort Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Diffuse Optical Spectroscopy Imaging - Neoadjuvant Chemo (NAC) Cohort: Diffuse Optical Spectroscopy Imaging (DOSI) at 6 time points.
  Interventions: Device: Diffuse Optical Spectroscopy Imaging (DOSI) - Neoadjuvant Chemo (NAC) Cohort
- Diffuse Optical Spectroscopy Imaging - Non-NAC Cohort: Diffuse Optical Spectroscopy Imaging (DOSI) at 1 time point.
  Interventions: Device: Diffuse Optical Spectroscopy Imaging (DOSI) - Non-NAC Cohort

INTERVENTIONS:
Device: Diffuse Optical Spectroscopy Imaging (DOSI) - Neoadjuvant Chemo (NAC) Cohort — Participants will have up to 9 DOSI scans at 6 different time points during the course of their neoadjuvant chemotherapy. The time course of chemotherapy may vary between 3-9 months depending on the type chemotherapy subjects receive. Depending on chemotherapy schedule, subjects may or may not be asked to participate in all the 6 measurement time points. The number of DOSI scans each subject requires will be decided during consent. Each DOSI scan will take about 30-60 minutes, although scans at infusion time point will take longer in total due to repeated or continuous measurements.
  Groups: Diffuse Optical Spectroscopy Imaging - Neoadjuvant Chemo (NAC) Cohort
Device: Diffuse Optical Spectroscopy Imaging (DOSI) - Non-NAC Cohort — Participants will have 1 DOSI scan at baseline. The DOSI scan will take about 30-60 minutes.
  Groups: Diffuse Optical Spectroscopy Imaging - Non-NAC Cohort

SUMMARY:
This study seeks to enroll women with breast cancer undergoing neoadjuvant chemotherapy to evaluate if Diffuse Optical Spectroscopy Imaging (DOSI) can predict a patient response to chemotherapy treatment. DOSI is a noninvasive imaging method that uses harmless near-infrared light using simple wearable probes held against the skin by transparent dressings to predict tumor metabolic activity. It uses nonionizing radiation, requires no external contrast agent and uses low light exposure to human tissue. DOSI scans can be performed frequently at the bedside in settings such as a doctor's office or infusion center.

DETAILED DESCRIPTION:
DOSI has already shown promise in monitoring breast cancer patients undergoing preoperative chemotherapy. Several groups have demonstrated optical changes predictive of response in the course of weeks to months of treatment. The investigators group has begun to show that DOSI measurements during drug infusions and at early time-points (first 24 hours) correlate with tumor final pathological response. While this data is provocative, significantly more work is needed to confirm that early time-points are predictive in different treatment groups and tumor molecular subtypes.

In this study, breast cancer patients will receive DOSI scans at a subset or all of the following time-points: baseline, during drug infusion, early therapy, mid-therapy and post-therapy. DOSI results will be compared to standard of care pathology results determined after surgery. Additionally, the investigators will correlate DOSI parameters with any additional biopsy specimens taken during treatment (typically for patients on adaptive treatment trials). Each DOSI scan will take about 30-60 minutes/ session, although infusion measurements will take longer. DOSI can potentially help doctors to gain information necessary to make evidence-based changes in treatment strategies of individual patients. The investigators long-term goal is to provide oncologists with a relatively simple, risk-free bedside tool that can help predict response early, thereby maximizing therapeutic response and minimizing unnecessary toxicity.

A cohort of 10 additional patients with breast cancer who are not receiving neoadjuvant chemotherapy (NAC) who will only be measured at baseline has been created. Complete characterization of baseline properties in patients is essential for understanding subsequent changes from baseline in response to chemotherapy. Adding an additional 10 patients who are not receiving NAC to be enrolled will allow for better characterization of baseline properties, which in turn will allow for a better understanding of the changes in properties seen in those patients who are undergoing NAC.

ELIGIBILITY:
Inclusion Criteria for Neoadjuvant Chemo (NAC) Cohort:

1. Female;
2. Diagnosis of invasive breast cancer by clinical breast examination, by standard of care diagnostic imaging, or by initial tissue biopsy;
3. Planned for primary systemic (neoadjuvant) chemotherapy and surgical resection of residual primary tumor following completion of neoadjuvant chemotherapy;
4. Tumor size ≥ 2cm, measured on imaging or estimated by physical exam;
5. Planned definitive breast surgery (mastectomy or lumpectomy/breast conservation) following completion of neoadjuvant therapy;
6. Age 18 years or older;
7. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2 (Karnofsky performance status ≥ 60%;
8. Adequate organ and marrow function, as defined at Boston Medical Center (BMC);
9. Postmenopausal for a minimum of one year, OR surgically sterile, OR not pregnant, confirmed by a pregnancy test as per institutional standard of care, and willing to use adequate contraception (hormonal or barrier method of birth control; abstinence) for the duration of study participation;
10. Able to understand and willing to sign a written informed consent document and a Health Insurance Portability and Accountability Act (HIPAA) authorization in accordance with institutional guidelines.

Inclusion Criteria for Non-NAC Cohort:

1. Female;
2. Diagnosis of invasive breast cancer by clinical breast examination, by standard of care diagnostic imaging, or by initial tissue biopsy;
3. Tumor size ≥2cm, measured on imaging or estimated by physical exam;
4. Planned definitive breast surgery (mastectomy or lumpectomy/breast conservation) following completion of neoadjuvant therapy;
5. Age 18 years or older;
6. ECOG Performance Status ≤ 2 (Karnofsky performance status ≥ 60%; see Appendix II);
7. Adequate organ and marrow function, as defined at BMC;
8. Postmenopausal for a minimum of one year, OR surgically sterile, OR not pregnant, confirmed by a pregnancy test as per institutional standard of care, and willing to use adequate contraception (hormonal or barrier method of birth control; abstinence) for the duration of study participation;
9. Able to understand and willing to sign a written informed consent document and a HIPAA authorization in accordance with institutional guidelines.

Exclusion Criteria for All Cohorts:

1. Previous treatment (chemotherapy, radiation, or surgery) to involved breast;
2. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements;
3. Medically unstable;
4. Under age 18;
5. Pregnant or nursing;
6. Previous malignancy, other than basal cell or squamous cell carcinoma of the skin or in situ carcinoma of the cervix, from which the patient has been disease free for less than 5 years;
7. No contraindications for primary chemotherapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The first cohort will consist of participants with up to 9 DOSI scans at 6 different time points during the course of their neoadjuvant chemotherapy (NAC). The time course of chemotherapy may vary between 3-9 months depending on the type chemotherapy subjects receive.
  There will be a second cohort of patients with breast cancer who are not receiving neoadjuvant chemotherapy (NAC) and who will only be measured at baseline.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2025-05-08 (Actual); Study Completion 2025-05-08 (Actual)

PRIMARY OUTCOMES:
Analysis of differences in longitudinal trends of oxyhemoglobin concentration as related to final pathological response | 6 months
  The longitudinal trends of oxyhemoglobin concentration measured over the early time-points (infusion, first 10 days). Differences in these trends will be analyzed to determine if they are prognostic of the final pathologic response (i.e. pathological complete response or non-complete response) of the primary tumor in patients with locally advanced breast cancer.

SECONDARY OUTCOMES:
Analysis of longitudinal trends of other composite DOSI derived parameters (deoxyhemoglobin, total blood volume, oxygen saturation, water, lips concentrations) | 6 months
  The longitudinal trends of other DOSI derived parameters (deoxyhemoglobin, total blood volume, oxygen saturation, water, lips concentrations) measured over the early time-points (infusion, first 10 days), mid therapy, and end therapy time-points.
Analysis of composite DOSI derived parameters (deoxyhemoglobin, total blood volume, oxygen saturation, water, lips concentrations) as related to overall pathologic response and to biopsy results | up to 6 months
  DOSI derived parameters (deoxyhemoglobin, total blood volume, oxygen saturation, water, lips concentrations) as measured immediately prior to a mid-therapy biopsy. These parameters will be correlated to overall pathologic response and to biopsy results.

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Ko, MD MPH, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-05-02): https://cdn.clinicaltrials.gov/large-docs/56/NCT02510456/ICF_000.pdf